CLINICAL TRIAL: NCT05098340
Title: Clinical Significance of Circulating circRNA in Acute Ischemic Stroke (CRAST)
Brief Title: Circulating circRNA in Acute Ischemic Stroke
Acronym: CRAST
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2021-KL107-01
Record Dates: First submitted 2021-10-17; First posted 2021-10-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
Keywords: circRNA
MeSH Terms: conditions — Ischemic Stroke | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — An 10 ml peripheral venous blood will be collected from the participants before and after interventions (i.e. intravenous thrombolysis and/or endovascular therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIS group: This group includes patients with acute ischemic stroke (AIS).
  Interventions: Genetic: Quantitative Real-time polymerase chain reaction
- HC group: This group includes healthy controls (HC).
  Interventions: Genetic: Quantitative Real-time polymerase chain reaction

INTERVENTIONS:
Genetic: Quantitative Real-time polymerase chain reaction — Quantitative Real-time polymerase chain reaction of circular RNA (circRNA).

SUMMARY:
CRAST is to analyze the expression pattern of circular RNA (circRNA) by bioinformatics analysis in patients with acute ischemic stroke and healthy control. The candidate circRNA will be verified as biomarkers for the detection and prognosis of acute ischemic stroke.

DETAILED DESCRIPTION:
Circular RNAs have been highlighted to be involved in the pathological process of ischemic stroke (IS). The purpose of this protocol will investigate the expression pattern of circular RNA (circRNA) by bioinformatics analysis in patients with acute ischemic stroke and healthy control. The candidate circRNA will be verified as biomarkers for the detection and prognosis of acute ischemic stroke. Distinctive expression patterns of circRNA will be identified by individual quantitative real time polymerase chain reaction (qRT-PCR). A diagnostic or predictive model will be established using logistic regression. The panel of these altered circRNAs may be associated with acute IS and could serve as a novel diagnostic or predictive method.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed acute ischemic stroke by a diffusion-weighted imaging-position lesion on magnetic resonance imaging (MRI) and a new lesion on a brain computed tomography (CT) scan
* Within 72 hours of symptom onset
* Good performance status
* Signed an approved informed consents

Exclusion Criteria:

* a history of hemorrhagic infarction, chronic kidney/liver diseases, peripheral arterial occlusive disease, active malignant disease, and inflammatory or infectious diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There will be 100 patients suspected of AIS (such as transient ischemic attack), 300 AIS patients and 100 Healthy controls，whose data will be applied for construction and validation of diagnostic and predictive models of circRNA from the circulating blood.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Differential expression pattern of circRNA | 90 days
  Differential expression pattern of circular RNA (circRNA) will be compared between AIS group and HC group, thus candidate circRNA will be verified as biomarkers for the detection and prognosis of AIS.

SECONDARY OUTCOMES:
Dynamic changes of circRNA during the follow-up period | 90 days
  Dynamic changes of circRNA will be explored before and after endovascular therapy
Correlation of circRNA and stroke-associated infection | 30 days
  Correlation of circRNA and stroke-associated infection will be explored in acute ischemic stroke.
Correlation of circRNA and inflammatory factors in acute ischemic stroke | 7 days
  Correlation of circRNA and inflammatory factors on admission will be explored in acute ischemic stroke.
Prognostic value of circRNA in acute ischemic stroke | 90 days
  The prognosis of AIS patients will be analyzed between differential expressed candidate circRNA after they have completed the systematic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No